CLINICAL TRIAL: NCT04348747
Title: A Phase IIa Study of Dendritic Cell Vaccines Against Her2/Her3 and Pembrolizumab in Patients With Asymptomatic Brain Metastasis From Triple Negative Breast Cancer (TNBC) or HER2+ Breast Cancer (HER2+BC) or Hormone Receptor Positive (HR+) Breast Cancer.
Brief Title: Dendritic Cell Vaccines Against Her2/Her3 and Pembrolizumab for the Treatment of Brain Metastasis From Triple Negative Breast Cancer or HER2+ Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-19-04120; NCI-2020-01520 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-19-04120 (Other: Roswell Park Cancer Institute); W81XWH-19-0674 (Other: DOD)
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Malignant Neoplasm in the Brain; Metastatic Triple-Negative Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Brain Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (anti-HER2/3 dendritic cell vaccine) (Experimental): TREATMENT PHASE: Patients receive anti-HER2/HER3 dendritic cell vaccine ID on days 1, 22, and 43. Patients will also receive pembrolizumab IV on the same days.
  MAINTENANCE PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients may also receive a booster dose of anti-HER2/3 dendritic cell vaccine ID, every 3-6 months in the opinion of principal investigator.
  Interventions: Biological: Anti-HER2/HER3 Dendritic Cell Vaccine; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Anti-HER2/HER3 Dendritic Cell Vaccine — Given ID
  Other Names: Anti-HER2/3 DC Vaccine; Anti-HER2/3 Dendritic Cell Vaccine
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase IIa trial studies how well dendritic cell vaccines against Her2/Her3 and pembrolizumab work for the treatment of triple negative breast cancer or HER2+ breast cancer or HER+ Breast cancer that has spread to the brain (brain metastasis). Dendritic cell vaccines work by boosting the immune system (a system in the body that protect against infection) to recognize and destroy the cancer cells. . Pembrolizumab is an "immune checkpoint inhibitor" which is designed to either "unleash" or "enhance" the cancer immune responses that already exist by either blocking inhibitory molecules" or by activating stimulatory molecules. Giving dendritic cell vaccines and pembrolizumab may shrink the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* I. The best overall central nervous system (CNS) response as per Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM).

SECONDARY OBJECTIVES:

* I. Volumetric quantification of brain metastases.
* II. The non-CNS (i.e. of systemic disease) response rate as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* III. The median CNS, non-CNS and overall progression free survival (PFS).
* IV. The median overall survival (OS).
* V. The safety of this regimen.
* VI. The proportion of patients not requiring retreatment for their brain metastasis at 6 months since the first dose of anti-HER2/3 vaccine.
* VII. Rate of failure of irradiated lesions.

OUTLINE:

TREATMENT PHASE: Patients receive anti-HER2/HER3 dendritic cell vaccine intradermally (ID) on days 1, 22, and 43. Patients also receive Pembrolizumab intravenous (IV) infusion on the same day.

MAINTENANCE PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients may also receive a booster dose of anti-HER2/HER3 dendritic cell vaccine ID, every 3-6 months in the opinion of principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* female participant is eligible to participate if she is not pregnant,not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP)
  * A WOCBP who agrees to follow contraceptive guidance
* WOCBP must agree to use acceptable birth control methods for the duration of the study and until persistence of the study drug is no longer detected in the peripheral blood:this may be a period of several years. Methods for acceptable birth control include: condoms, diaphragm or cervical cap with spermicide, intrauterine device, and hormonal contraception; it is recommended that a combination of two methods be used. NOTE: If the risk of conception exists, patients must agree to use highly effective contraception throughout the study and for at least two years following the last study treatment administration
* Negative serum and highly sensitive urine pregnancy test(s):

  i) within 72 hours prior to study allocation; ii) following initiation of treatment, pregnancy testing will be performed for WOCBP and interpreted prior to every cycle of pembrolizumab (Initial Treatment Phase); iii) at the End of Treatment (EOT) Assessment; and iv) whenever pregnancy is otherwise suspected. Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test must be performed and must be negative in order for subject to start receiving study medication.
* Histologically or cytologically confirmed diagnosis of triple negative breast cancer (TNBC) (estrogen receptor [ER] =< 1%, progesterone receptor [PR] =< 1% HER2 negative) or HR+ breast cancer

  * HER2 testing should be performed on the invasive component using a validated immunohistochemistry (IHC) or in situ hybridization (ISH) assay
  * IHC staining is defined as:

    * IHC 3+ if there is complete and intense circumferential membrane staining within > 10 percent of tumor cells. All IHC 3+ tumors are considered HER2 positive
    * IHC 2+ if there is incomplete and/or weak/moderate, circumferential membrane staining within > 10 percent of tumor cells. All IHC 2+ tumors are reported as HER2 equivocal
    * IHC 1+ if there is faint or barely perceptible, incomplete membrane staining within > 10 percent of tumor cells. All IHC 1+ tumors are reported as HER2 negative
    * IHC 0 if (1) no staining is observed, or (2) there is faint or barely perceptible, incomplete membrane staining within < 10 percent of tumor cells. All IHC 0 tumors are reported as HER2 negative
    * Equivocal HER2 testing should trigger reflex HER2 testing using ISH on the same specimen or a new test (using a different specimen with either IHC or ISH)
  * Results from ISH are defined as the ratio of gene amplification of HER2 and the chromosome 17 enumeration probe (CEP17). Results are reported as:

    * ISH positive if the HER2/CEP17 ratio is >= 2.0, and the HER2 copy number signals/cell is >= 4
    * Definitive diagnosis will be rendered pending further workup in the following instances:

      * If the HER2/CEP17 ratio is >= 2.0 and an average HER2 copy number is < 4.0 signals/cell - negative if confirmed on retesting
      * If the HER2/CEP17 ratio is < 2.0 and the average HER2 copy number is >= 6.0 signals/cell positive - if confirmed on retesting
      * If the HER2/CEP17 ratio is < 2.0 and an average HER2 copy number is between >= 4.0 and < 6.0 signals/cell negative - if confirmed on retesting
    * ISH negative if the HER2/CEP17 ratio is < 2.0 and average HER2 copy number is < 4.0 signals/cell
* Measurable brain disease as per RANO-BM criteria modified to include the cut off point of 0.5 cm or higher. Have at least one untreated (includes irradiation) brain metastasis approved by a research team that meets the following size requirements:

  * >= 0.5 cm AND twice the magnetic resonance imaging (MRI) slice thickness; and
  * < 3.0 cm, that is asymptomatic and does not require local therapy at the time of enrollment (i.e. target lesion[s])
  * Of note, lesions >= 0.5 cm and < 3 cm may be determined ineligible by the research team because of location or symptoms. An untreated brain metastasis is defined as a lesion not present at the time of whole brain radiation therapy or not included in a stereotactic radiotherapy field (or within 0.5 cm of a treated lesion), or any lesion that is new or unequivocally progressing since prior radiation therapy or prior surgery.
* Any brain metastasis >= 3.0 cm or causing symptoms must have previously been treated with local therapy (i.e. radiation or surgical resection, as clinically appropriate) prior to study enrollment. Any lesion present at the time of whole brain radiation therapy (WBRT) or included in the stereotactic radiotherapy field (or within 5 mm of the treated lesion) will NOT be considered evaluable unless it is new or documented to have progressed since treatment
* Stereotactic radiosurgery (SRS) and/or prior radiotherapy is permitted >=2 weeks prior to initial Dendritic Cell (DC) vaccine dose (leaving one or more lesions which are not radiated and will be used as target lesions) but a follow up brain MRI should be obtained prior to dendritic cell (DC) vaccine to determine stability of the lesions. An interval of at least 4 weeks after the end of whole brain radiation or for any surgical resection of brain lesions is permitted ; an interval of at least 4 weeks or 5 half-lives (whichever is sorter) after the last cytotoxic, targeted, immunotherapeutic or investigational agent is permitted (prior to the start of DC vaccine)

  * Previous whole brain radiation is allowed if patient has been diagnosed with recurrent, progressive brain metastasis. Previously irradiated lesions would be considered non-target lesions
  * Previously resected lesions or those treated with SRS would be considered nontarget lesions. There is no limitation on prior local therapies to other lesions.
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Toxicity that has not recovered to <=Grade 1 is allowed if it meets the inclusion requirments for lab parameters (Participants with <= Grade 2 neuropathy may be eligible)
* Patients must have adequate organ and marrow function as defined below (specimens must be collected within 10 days prior to the start of study treatment):
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L
* Leukocytes: >= 3 x 10^9/L
* Absolute neutrophil count: >= 1.5 x 10^9/L
* Platelets: >= 100 x 10^9/L
* Total bilirubin: =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): =< 2.5 x institutional upper limit of normal (=< 5 x ULN for participants with liver metastases)
* Creatinine OR Measured or calculated creatinine clearance (Glomerular Filtration Rate (GFR) can also be used in place of creatinine or CrCl): ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
* International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (APTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* No evidence of leptomeningeal disease
* If patient is on steroids, they must be on a steroid dose less than or = to an equivalent prednisone dose of 10 mg daily
* Life expectancy of > 3 months
* Prior checkpoint inhibitors permitted 3 weeks prior to enrollment
* If the disease has progressed on current treatment in the CNS, prior to consent, patients may continue Her 2 directed antibody treatment (trastuzumab and pertuzumab); aromatase inhibitor or tamoxifen while on the study; patients with triple negative breast cancer may continue capecitabine, eribulin or paclitaxel while on study per PI discretion
* Patients with systemic disease will be managed as detailed in Section 10.1 - Patients who develop systemic disease progression on the protocol will be managed as detailed in Section 10.4.2

Exclusion Criteria:

* Any condition which might confound the results of the study, interfere with the subject's participation for full participation (for the full duration of the study) or in the Investigator's opinion deems the participant an unsuitable candidate for the study
* Symptomatic brain metastases. Any neurologic symptoms present must have resolved with local therapy by the time of administration of study drugs
* May not be receiving any other investigational agents and may not have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of DC vaccine treatment
* Has had prior chemotherapy or targeted small molecule therapy (except treatment mentioned in inclusion criteria 17) within 4 weeks or 5 half-lives (whichever is sooner) prior to start of treatment (first DC vaccine) or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent. Previous radiation to extracranial sites may be completed at any time prior to initiation of study drugs (first DC vaccine) with a 2-week washout is required.
* Rapidly progressing systemic disease which might interfere with completion of all the vaccine doses
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* History of allogenic tissue/solid organ transplantation
* Has an active infection requiring systemic therapy which in the investigator's opinion will increase risk to the patient
* Has known active hepatitis B or hepatitis C infection (Testing is not mandatory)
* Has known immunosuppressive disease (e.g. human immunodeficiency virus [HIV], acquired immunodeficiency syndrome [AIDS] or other immune depressing disease). Testing is not mandatory
* Has received a blood transfusion in the two weeks prior to leukapheresis
* Pregnant or actively nursing (females who agree to stop nursing would be eligible) participants
* Unwilling or unable to follow protocol requirements
* Brain lesion size with significant midline shift or obstructive hydrocephalus
* The use of corticosteroids to control cerebral edema or treat neurologic symptoms will not be allowed unless at a low dose, not to exceed 10 mg of prednisone (or equivalent) per day
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* History of (non-infectious) pneumonitis /interstitial lung disease that required steroids, or has current pneumonitis/ interstitial lung disease
* Presence of leptomeningeal disease
* Any contraindication to MRI (i.e., patients with pacemakers or other metal implanted medical devices). An MRI safety questionnaire is required prior to MR imaging
* Has received prior radiotherapy within 2 weeks of start of study treatment with dendritic cell (DC) vaccine and/or has received SRS <2. weeks prior to the administration of the first DC vaccine dose. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-CNS disease
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Seasonal influenza vaccines for injection are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed. Administration of killed vaccines is allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug (DC vaccine)
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* A WOCBP who has a positive urine or blood pregnancy test within 72 hrs prior to study allocation.

  *Note: in the event that 72 hrs have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
* Known active carcinomatous meningitis
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Central nervous system (CNS) objective response rate (ORR) | Up to 2 years
  Assessed per Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) working group. Will be summarized using frequencies and relative frequencies. A 90% confidence interval about the true ORR will be obtained using Jeffrey's prior method.

SECONDARY OUTCOMES:
Volumetric quantification of brain metastases | Up to 2 years
Non-CNS (i.e. of systemic disease) response rate | Up to 2 years
  Assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Median CNS progression free survival (PFS) | Up to 2 years
  Will be summarized using frequencies and relative frequencies. A 90% confidence interval about the true response rate will be obtained using Jeffrey's prior method.
Non-CNS PFS | Up to 2 years
  Will be summarized using frequencies and relative frequencies. A 90% confidence interval about the true response rate will be obtained using Jeffrey's prior method.
Overall PFS | Up to 2 years
  Will be summarized using frequencies and relative frequencies. A 90% confidence interval about the true response rate will be obtained using Jeffrey's prior method.
Proportion of patients who have a CNS PFS | At 6 months
Median overall survival (OS) | Up to 2 years
Incidence of adverse events | Up to 2 years
  Safety of the regimen characterized by type, frequency, severity (according to Common Terminology Criteria for Adverse Events [CTCAE] version 5.0), timing, seriousness and relationship to study treatment. All toxicities and adverse events will be summarized by grade using frequencies and relative frequencies.
Proportion of patients not requiring retreatment for their brain metastasis at 6 months since the first dose of anti-HER2/3 vaccine | At 6 months
  Will be summarized using standard Kaplan-Meier methods. Estimates of the median time and 6-month rates will be obtained with 90% confidence intervals.
Rate of failure of irradiated lesions | Up to 2 years

OTHER OUTCOMES:
Changes in tumor circulating tumor lymphocyte (CTL)s | Baseline up to 2 years
  Will be summarized by timepoint using the mean and standard deviation; and graphically using box- or dot-plots. The mean change (pre- to post-treatment) in biomarker values will be evaluated using a two-sided, permutation paired t-tests. The correlation between different biomarkers or changes in biomarkers will be evaluated using the Spearman correlation coefficient. The association between biomarker values (baseline or change) and response will be evaluated using logistic regression models.
Changes in tumor PDL-1 expression | Baseline up to 2 years
  Will be summarized by timepoint using the mean and standard deviation; and graphically using box- or dot-plots. The mean change (pre- to post-treatment) in biomarker values will be evaluated using a two-sided, permutation paired t-tests. The correlation between different biomarkers or changes in biomarkers will be evaluated using the Spearman correlation coefficient. The association between biomarker values (baseline or change) and response will be evaluated using logistic regression models.
Changes in cytokine expression | Baseline up to 2 years
  Will be summarized by timepoint using the mean and standard deviation; and graphically using box- or dot-plots. The mean change (pre- to post-treatment) in biomarker values will be evaluated using a two-sided, permutation paired t-tests. The correlation between different biomarkers or changes in biomarkers will be evaluated using the Spearman correlation coefficient. The association between biomarker values (baseline or change) and response will be evaluated using logistic regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Sheheryar Kabraji, BMBCh, Principal Investigator — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia